CLINICAL TRIAL: NCT07162311
Title: Effect of Home-Based Transcranial Direct Current Stimulation on Pain in Patients With Rheumatoid Arthritis With Low Inflammatory Activity: A Randomized, Double-Blind, Sham-Controlled Clinical Trial
Brief Title: Effect of Home-Based Transcranial Direct Current Stimulation on Pain in Patients With Rheumatoid Arthritis With Low Inflammatory Activity
Acronym: tDCS RA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Stephanie Pilotti, Principal Investigator; PhD Student in Medical Sciences at the Federal University of Rio Grande do Sul, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-0014
Record Dates: First submitted 2025-04-07; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-04

CONDITIONS: Rheumatic Arthritis; Chronic Pain
Keywords: Rheumatoid arthrtis; chronic pain; tDCS
MeSH Terms: conditions — Rheumatic Fever; Chronic Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acitve tDCS (Active Comparator): 2 mA, 20 minutes/day, 5 days/week, for 4 weeks, applied at home under remote supervision.
  Interventions: Device: tDCS
- Sham tDCS (Sham Comparator): Same parameters as active tDCS, but current was ramped down after 30 seconds to mimic sensation without delivering stimulation.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Home-Based Transcranial Direct Current Stimulation

SUMMARY:
Rheumatoid arthritis (RA) is a highly complex inflammatory autoimmune disease. Several drugs have been developed in recent decades to target the immune components of inflammation. However, even with effective anti-inflammatory and immunosuppressive therapies for controlling RA, many patients still report significant levels of chronic pain due to CNS neuroplasticity, perpetuating physical disability, psychosocial problems, decreased work activity, and poor quality of life. In addition, chronic pain can lead to increased public spending due to the need for more medical visits, ineffective drug treatments, and financial disability benefits. Transcranial stimulation (a noninvasive neural stimulation technique with minimal adverse effects and easy home use) has been a promising adjunct tool in the treatment of chronic pain and psychological disorders in diseases that affect the central nervous system in the long term. Thus, exploring transcranial direct current stimulation in RA patients with low levels of inflammation could impact on improving pain, functionality, psychological aspects and overall quality of life, as well as reducing healthcare costs for society.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a highly complex inflammatory autoimmune disease. Several drugs have been developed in recent decades to target the immune components of inflammation. However, even with effective anti-inflammatory and immunosuppressive therapies for controlling RA, many patients still report significant levels of chronic pain due to CNS neuroplasticity, perpetuating physical disability, psychosocial problems, decreased work activity, and poor quality of life. In addition, chronic pain can lead to increased public spending due to the need for more medical visits, ineffective drug treatments, and financial disability benefits. Transcranial stimulation (a noninvasive neural stimulation technique with minimal adverse effects and easy home use) has been a promising adjunct tool in the treatment of chronic pain and psychological disorders in diseases that affect the central nervous system in the long term. Thus, exploring transcranial direct current stimulation in RA patients with low levels of inflammation could impact on improving pain, functionality, psychological aspects and overall quality of life, as well as reducing healthcare costs for society.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18-70 with RA.
* Participants with generalized pain ≥ 40 mm on the VAS-Pain scale, lasting over 3 months, and not of mechanical or inflammatory origin, as assessed by a certified rheumatologist.
* Evidence of low inflammatory markers, including with C-reactive protein (CRP) <10 mg/dL and sedimentation rate (ESR) <20 mm/h, and stable treatment for PsA for at least 6 months prior to study enrollment.

Exclusion Criteria:

* History of brain surgery, traumatic brain injury, stroke, previous intracranial metal implantation, pregnancy, or breastfeeding.
* Previous history of autoimmune diseases other than RA.
* History of neurological diseases.
* Previous history of neoplasia.
* History of any other uncompensated clinical disease.
* Use of illicit drugs within the past 6 months.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-12-22 (Estimated); Study Completion 2028-12-22 (Estimated)

PRIMARY OUTCOMES:
VAS pain | Visual Analog Scale (VAS, 0-100 mm; higher scores indicate worse pain) assessed at baseline (Day 1), after 10 days of tDCS treatment, at Week 4 of tDCS treatment (end of treatment), and at 3, 6, 9, and 12 months post-treatment.
  Visual Analogue Scale for pain

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No
The Individual Patient Data (IPD) will not be shared due to privacy and confidentiality concerns, as well as the protection of sensitive patient information. Additionally, there may be legal or regulatory restrictions that prevent the release of such data. Sharing of IPD could also raise ethical issues regarding informed consent and the use of data beyond the initial scope of the study.

REFERENCES:
- [Background] Caumo W, Lopes Ramos R, Vicuna Serrano P, da Silveira Alves CF, Medeiros L, Ramalho L, Tomeddi R, Bruck S, Boher L, Sanches PRS, Silva DP Jr, Ls Torres I, Fregni F. Efficacy of Home-Based Transcranial Direct Current Stimulation Over the Primary Motor Cortex and Dorsolateral Prefrontal Cortex in the Disability Due to Pain in Fibromyalgia: A Factorial Sham-Randomized Clinical Study. J Pain. 2024 Feb;25(2):376-392. doi: 10.1016/j.jpain.2023.09.001. Epub 2023 Sep 7. PMID 37689323